CLINICAL TRIAL: NCT05920720
Title: Personalizing Disordered Eating Treatment Using Mobile Technology: Self-Guided, Personalized Treatment for Women
Brief Title: Self-Guided Personalized Treatment for Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Cheri Levinson, Director, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#23.0274; 5P20GM103436-23 (NIH)
Record Dates: First submitted 2023-06-09; First posted 2023-06-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Disordered Eating
Keywords: Treatment; Therapy; Anorexia Nervosa; Bulimia Nervosa; Binge Eating Disorder; Atypical Anorexia Nervosa; Other specified feeding and eating disorder
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-guided Personalized Treatment (Experimental): Women who endorse significant DE will complete two weeks of smart-phone self-monitoring to identify target problems and will be sent two self-guided modules of personalized treatment directly to their smart-phones.
  Interventions: Behavioral: Self-guided Personalized Treatment

INTERVENTIONS:
Behavioral: Self-guided Personalized Treatment — Women who endorse significant DE will complete two weeks of smart-phone self-monitoring to identify target problems and will be sent two self-guided modules of personalized treatment directly to their smart-phones.
  Other Names: Personalized Treatment

SUMMARY:
The investigators plan to collect preliminary data on the feasibility, acceptability, and user uptake of a personalized self-guided mobile intervention for disordered eating (DE) and test the initial clinical efficacy of this intervention. Women (N=50) who endorse significant DE will complete two weeks of smart-phone self-monitoring to identify target problems and will be sent two self-guided modules of personalized treatment directly to their smart-phones. The investigators will assess engagement with the modules throughout two months and administer baseline, week 5, and week 8 assessments for acceptability, uptake, and initial clinical efficacy (e.g., DE symptoms, anxiety, quality of life). The investigators will also complete a focus group (n=10) with a subset of users to receive input on the mobile-application assessment and ease of self-guided intervention modules.

ELIGIBILITY:
Inclusion Criteria:

* Endorse disordered eating (score of 2.3 or above on EDE-Q6)
* Age 18-65
* Ability to read and write English
* Own a smartphone or tablet

Exclusion Criteria:

* Active mania
* Active suicidality
* Active psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will be self-identified women.
Enrollment: 50 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Disordered eating symptoms | Up to 8 weeks
  Changes in disordered eating symptoms will be assessed with the Eating Disorder Examination Questionnaire-6 (EDE-Q6)
Anxiety | Up to 8 weeks
  Changes in anxiety will be assessed with the Penn State Worry Questionnaire (PSWQ)
Depression | Up to 8 weeks
  Changes in depression will be assessed with the Beck Depression Inventory-2 (BDI-2)
Clinical Impairment | Up to 8 weeks
  Changes in clinical impairment will be assessed with the Clinical Impairment Assessment (CIA)
Quality of life | Up to 8 weeks
  Changes in quality of life will be assessed with the Quality of Life Scale (QOLS)

CONTACTS AND LOCATIONS:
Overall Officials: Cheri A Levinson, Principal Investigator — University of Louisville
Locations (1):
- Eating Anxiety Treatment Laboratory and Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levinson CA, Williams BM, Christian C, Hunt RA, Keshishian AC, Brosof LC, Vanzhula IA, Davis GG, Brown ML, Bridges-Curry Z, Sandoval-Araujo LE, Ralph-Nearman C. Personalizing eating disorder treatment using idiographic models: An open series trial. J Consult Clin Psychol. 2023 Jan;91(1):14-28. doi: 10.1037/ccp0000785. PMID 36729494
- [Background] Borsboom D, Cramer AO. Network analysis: an integrative approach to the structure of psychopathology. Annu Rev Clin Psychol. 2013;9:91-121. doi: 10.1146/annurev-clinpsy-050212-185608. PMID 23537483
- [Background] Levinson CA, Hunt RA, Keshishian AC, Brown ML, Vanzhula I, Christian C, Brosof LC, Williams BM. Using individual networks to identify treatment targets for eating disorder treatment: a proof-of-concept study and initial data. J Eat Disord. 2021 Nov 4;9(1):147. doi: 10.1186/s40337-021-00504-7. PMID 34736538